CLINICAL TRIAL: NCT04042519
Title: The Correlation Research Between the Omega-3 and Omega-6 Inflammatory Metabolites and Stable COPD.
Brief Title: The Research of Metabolomics on COPD
Acronym: COPD
Status: Completed | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: The Fifth Affiliated Hospital of Zunyi Medical College (Other)
Responsible Party: Principal Investigator, LuQian Zhou, Associate professor of respiratory medicine, Guangzhou Institute of Respiratory Disease
Other Study IDs: MG-201909
Record Dates: First submitted 2019-07-29; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Metabolomics; Omega 6; Omega 3; COPD
Keywords: Metabolomics; Omega 6; Omega 3; COPD; lung function tests
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Healthy control: age - and sex-matched healthy individuals without lung disease
  Interventions: Diagnostic Test: Routine blood test
- Patients with mild and moderate COPD: Grading according to the GOLD guide standards
  Interventions: Diagnostic Test: Lung function test was performed on the subjects with Jaeger lung function instrument of Germany.; Diagnostic Test: Agilent 1290 Infinity LC system (UHPLC, Santa Clara CA) was used for Targeted metabolite detection.; Diagnostic Test: Routine blood test
- Patients with severe and very severe COPD: Grading according to the GOLD guide standards
  Interventions: Diagnostic Test: Lung function test was performed on the subjects with Jaeger lung function instrument of Germany.; Diagnostic Test: Agilent 1290 Infinity LC system (UHPLC, Santa Clara CA) was used for Targeted metabolite detection.; Diagnostic Test: Routine blood test
- The severe and very severe COPD group baseline: Severe and very severe COPD patients were in the baseline time group
  Interventions: Diagnostic Test: Lung function test was performed on the subjects with Jaeger lung function instrument of Germany.; Diagnostic Test: Agilent 1290 Infinity LC system (UHPLC, Santa Clara CA) was used for Targeted metabolite detection.; Diagnostic Test: Routine blood test
- The severe and very severe COPD group six months: Patients with severe and very severe COPD were six months from baseline.
  Interventions: Diagnostic Test: Lung function test was performed on the subjects with Jaeger lung function instrument of Germany.; Diagnostic Test: Agilent 1290 Infinity LC system (UHPLC, Santa Clara CA) was used for Targeted metabolite detection.; Diagnostic Test: Routine blood test
- The severe and very severe COPD group one year: Patients with severe and very severe COPD were one year from baseline.
  Interventions: Diagnostic Test: Lung function test was performed on the subjects with Jaeger lung function instrument of Germany.; Diagnostic Test: Agilent 1290 Infinity LC system (UHPLC, Santa Clara CA) was used for Targeted metabolite detection.; Diagnostic Test: Routine blood test

INTERVENTIONS:
Diagnostic Test: Lung function test was performed on the subjects with Jaeger lung function instrument of Germany. — This Jaeger lung function instrument of Germany is used to test the pulmonary ventilation function of COPD patients. Since the condition requires drug control and treatment, the drug cannot be stopped.
  Groups: Patients with mild and moderate COPD; Patients with severe and very severe COPD; The severe and very severe COPD group baseline; The severe and very severe COPD group one year; The severe and very severe COPD group six months
Diagnostic Test: Agilent 1290 Infinity LC system (UHPLC, Santa Clara CA) was used for Targeted metabolite detection. — We used the Agilent 1290 Infinity LC system mass spectrometer to analyze and detect metabolite peaks of patients according to retention time and mass/charge ratio after preliminary experiments and derivatization.
  Groups: Patients with mild and moderate COPD; Patients with severe and very severe COPD; The severe and very severe COPD group baseline; The severe and very severe COPD group one year; The severe and very severe COPD group six months
Diagnostic Test: Routine blood test — Blood routine test results include CRP, PCT, white blood cell count, red blood cell count, neutrophil percentage, eosinophil, basophil, et al.

SUMMARY:
Targeted metabolomics research was conducted on patients with chronic obstructive pulmonary disease (COPD). The correlation analyst between inflammation-related metabolites and lung function was analyzed by explored the metabolic pathways of inflammation-related omega-6 and omega-3 and combining them with lung function.

DETAILED DESCRIPTION:
Based on the global initiative for chronic obstructive pulmonary disease, the 80 confirmed stable COPD patients with mild-to-moderate were involved, 80 COPD patients with severe and very severe, and age, sex, all matching 40 cases without lung disease. The participants information was collected. Whole blood and pulmonary function were examined at three time points: admission, six months and one year, at the same time, targeted metabolomic analysis method are applied to detect serum metabolites, According to the access to assess the different severity of COPD in the stable period and the level of metabolites in different admission periods. After that, correlation analysis was conducted with pulmonary function indicators and other clinical indicators to observe the research value of inflammation-related metabolites in the development of COPD.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis
* The age ranges from 40 to 80
* No other pulmonary diseases
* No immune-related diseases

Exclusion Criteria:

* Not consistent with COPD diagnosis
* Age is out of range
* Interstitial lung disease, asthma and other lung diseases
* Immune system diseases
* Lost to follow-up

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Based on the global initiative for chronic obstructive pulmonary disease, the 80 confirmed stable COPD patients with mild-to-moderate were involved, 80 COPD patients with severe and very severe, and age, sex, all matching 40 cases without lung disease. The participants information was collected. Whole blood and pulmonary function were examined at three time points: admission, six months and one year, at the same time, targeted metabolomic analysis method are applied to detect serum metabolites, According to the access to assess the different severity of COPD in the stable period and the level of metabolites in different admission periods.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | October 1, 2016 to October 1, 2018
  The FEV1 percentage of predicted value is an important indicator in the diagnosis and treatment of COPD, and plays an important role in the severity rating.
  * level (mild) : FEV1 / FVC < 70%, FEV1% pred > 80%. Ⅱ level (moderate) : FEV1 / FVC < 70%, 50% ≦ FEV1% pred< 80%. Ⅲ level (severe) : FEV1 / FVC < 70%, 30% ≦ FEV1% pred < 50%. IV level (very severe) : FEV1/FVC<70%, FEV1% pred < 30%, or FEV1% pred <50% with chronic respiratory failure.
Forced vital capacity (FVC) | October 1, 2016 to October 1, 2018
  FVC is an important index to determine the resistance of respiratory tract. FEV1 and FEV1/FVC% in patients with obstructive airway obstruction, such as patients with chronic obstructive pulmonary disease, were reduced due to airway obstruction and prolonged expiratory.
FEV1/FVC ratio | October 1, 2016 to October 1, 2018
  This index is an important basis for the diagnosis of COPD and is crucial in the early stage of the disease to the later stage of the evaluation.
The metabolites of Omega-6 inflammatory indicator | October 1, 2016 to October 1, 2018
  Agilent 1290 Infinity LC system (UHPLC, Santa Clara CA) was used for the targeted determination of metabolites in the serum of subjects.
  Omega6 metabolites are closely related to inflammation and have been shown to be involved in a variety of diseases such as COPD, rheumatism, cardiovascular disease, et al.
The metabolites of Omega-3 inflammatory indicator | October 1, 2016 to October 1, 2018
  As an important anti-inflammatory factor, omega-3 is widely used in chronic inflammatory diseases, which can fight against the pro-inflammatory metabolites of omega-6.

SECONDARY OUTCOMES:
C-reaction protein | October 1, 2016 to October 1, 2018
  CRP is an acute phase protein synthesized by liver cells in response to inflammatory stimuli such as microbial invasion or tissue injury. Can reflect the inflammation level in COPD patients.
Leukocyte Count | October 1, 2016 to October 1, 2018
  White blood cells are very important blood cells in human blood. White blood cells bear many important tasks in the human body. They have the function of swallowing foreign bodies and producing antibodies.

IPD SHARING:
Plan to Share IPD: Yes
In this study, smoking time data were also included. Next, we plan to grade smoking time or sick time(Time from baseline or from the time of first diagnosis) to evaluate the change trend of inflammation-related metabolites.
Supporting Information: SAP
Time Frame: We will use the part of data for smoking-related research projects until 2020-06-01.
Access Criteria: Patients aged 40 to 80 diagnosed with stable COPD according to diagnostic criteria were selected, regardless of gender. No lung tumor, no interstitial lung disease, no immune-related lung disease. The patient himself or his family signed the informed consent for the experiment.

REFERENCES:
- [Background] Das UN. Ageing: Is there a role for arachidonic acid and other bioactive lipids? A review. J Adv Res. 2018 Feb 15;11:67-79. doi: 10.1016/j.jare.2018.02.004. eCollection 2018 May. PMID 30034877
- [Background] Serkova NJ, Standiford TJ, Stringer KA. The emerging field of quantitative blood metabolomics for biomarker discovery in critical illnesses. Am J Respir Crit Care Med. 2011 Sep 15;184(6):647-55. doi: 10.1164/rccm.201103-0474CI. Epub 2011 Jun 16. PMID 21680948
- [Background] Fulton AS, Hill AM, Williams MT, Howe PR, Frith PA, Wood LG, Garg ML, Coates AM. Feasibility of omega-3 fatty acid supplementation as an adjunct therapy for people with chronic obstructive pulmonary disease: study protocol for a randomized controlled trial. Trials. 2013 Apr 24;14:107. doi: 10.1186/1745-6215-14-107. PMID 23782589
- [Background] Tantucci C, Modina D. Lung function decline in COPD. Int J Chron Obstruct Pulmon Dis. 2012;7:95-9. doi: 10.2147/COPD.S27480. Epub 2012 Feb 9. PMID 22371650
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] D'Archivio M, Scazzocchio B, Giammarioli S, Fiani ML, Vari R, Santangelo C, Veneziani A, Iacovelli A, Giovannini C, Gessani S, Masella R. omega3-PUFAs exert anti-inflammatory activity in visceral adipocytes from colorectal cancer patients. PLoS One. 2013 Oct 7;8(10):e77432. doi: 10.1371/journal.pone.0077432. eCollection 2013. PMID 24116229
- [Background] Lemoine S CM, Brigham EP, Woo H, Hanson CK, McCormack MC, Koch A, Putcha N, Hansel NN. Omega-3 fatty acid intake and prevalent respiratory symptoms among U.S. adults with COPD. BMC Pulm Med. 2019 May 21;19(1):97. doi: 10.1186/s12890-019-0852-4. PMID 31122230
- [Background] Kilk K, Aug A, Ottas A, Soomets U, Altraja S, Altraja A. Phenotyping of Chronic Obstructive Pulmonary Disease Based on the Integration of Metabolomes and Clinical Characteristics. Int J Mol Sci. 2018 Feb 27;19(3):666. doi: 10.3390/ijms19030666. PMID 29495451
- [Background] Wang Y, Xu J, Meng Y, Adcock IM, Yao X. Role of inflammatory cells in airway remodeling in COPD. Int J Chron Obstruct Pulmon Dis. 2018 Oct 12;13:3341-3348. doi: 10.2147/COPD.S176122. eCollection 2018. PMID 30349237
- [Background] Pizzini A, Lunger L, Sonnweber T, Weiss G, Tancevski I. The Role of Omega-3 Fatty Acids in the Setting of Coronary Artery Disease and COPD: A Review. Nutrients. 2018 Dec 2;10(12):1864. doi: 10.3390/nu10121864. PMID 30513804
- [Background] Mesaros C, Blair IA. Targeted chiral analysis of bioactive arachidonic Acid metabolites using liquid-chromatography-mass spectrometry. Metabolites. 2012 Apr 20;2(2):337-65. doi: 10.3390/metabo2020337. PMID 24957514
- [Background] Schrimpe-Rutledge AC, Codreanu SG, Sherrod SD, McLean JA. Untargeted Metabolomics Strategies-Challenges and Emerging Directions. J Am Soc Mass Spectrom. 2016 Dec;27(12):1897-1905. doi: 10.1007/s13361-016-1469-y. Epub 2016 Sep 13. PMID 27624161